CLINICAL TRIAL: NCT03881033
Title: Determination of Optimal Mask Ventilation Mode in Pediatrics Using Real-time Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-18-192
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Ventilator Lung; Ultrasound

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P12 (Placebo Comparator)
  Interventions: Other: Peak inspiratory pressure
- P7+5 (Active Comparator)
  Interventions: Other: Peep 5cmH2O

INTERVENTIONS:
Other: Peep 5cmH2O — Face mask ventilation with peak inspiratory pressure according to the group P7+5 means face mask ventilation with peak inspiratory pressure 7cmH2O plus PEEP 5 cmH2O.
  Other Names: Peak inspiratory pressure
  Arms: P7+5
Other: Peak inspiratory pressure — Face mask ventilation with peak inspiratory pressure according to the group P12 means face mask ventilation with peak inspiratory pressure 12cmH2O without PEEP.
  Arms: P12

SUMMARY:
The peak inspiratory pressure during face mask ventilation for general anesthesia is closely correlated with gastric insufflation. High pressure increases the amount of air in stomach and low pressure could decrease the tidal volume, therefore ideal pressure means the pressure guarantee adequate ventilation with minimal gastric insufflation.

The aim of this study is finding the proper pressure and mode of face mask ventilation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* The ASA class I,II and 1-5 years pediatric patients need general anesthesia

Exclusion Criteria:

* Oropharyngeal or facial pathology accompanied
* Obese (BMI > 30 kg/m2)
* GI tract obstruction

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
The degree of atelectasis | 1min after ventilator-on
  After intubation, confirming endotracheal intubation, the ventilator is connected and turned on.

SECONDARY OUTCOMES:
The incidence of gastric insufflation | During face mask ventilation